CLINICAL TRIAL: NCT05187000
Title: Effect of Individualized Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Disorder of Consciousness
Brief Title: Effects of Individualized rTMS in DOC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qiuyou Xie (Other)
Responsible Party: Sponsor-Investigator, Qiuyou Xie, principal investigator, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L20210505
Record Dates: First submitted 2021-11-26; First posted 2022-01-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Disorder of Consciousness; Transcranial Magnetic Stimulation
Keywords: Disorder of Consciousness; repetitive transcranial magnetic stimulation; randomized control trial
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Stimulation Group for Cross Study (Sham Comparator): Sham stimulation will be delivered on the patients head using a sham coil in the crossover study.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation
- Individualized rTMS Group for Cross Study (Experimental): Real stimulation will be delivered on individualized target using a real coil in the crossover study.
  Interventions: Device: individualized repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: individualized repetitive transcranial magnetic stimulation — During the rTMS-active stage, treatment will be given for 10 consecutive sessions (one session daily). The participants will be placed in the semi-reclining position on either a normal chair or a wheelchair and each stimulation session will last 20 minutes with a frequency of 10 Hz (train duration: 1s; inter-train interval: 5s; 200 effective stimulation series; 2000 pulses at 90% of RMT).
  Arms: Individualized rTMS Group for Cross Study
Device: Sham repetitive transcranial magnetic stimulation — The sham coil will be used which has no magnetic field to send to the cerebral cortex while appearing to be the same shape as the active coil, with good approximation of auditory feedback.
  Arms: Sham Stimulation Group for Cross Study

SUMMARY:
Background: Disorder of consciousness(DOC) is a series of arousal and cognitive disorders secondary to the most severe brain injury. Once a patient is diagnosed with a DOC, a poor prognosis is assumed and the rehabilitation for whom is greatly limited. Therefore, the treatment of DOC poses extraordinary challenges. Various treatments protocols have been reported of successful in promoting rehabilitation of DOC patients. Repetitive transcranial magnetic stimulation(rTMS), as a non-invasive brain stimulation technique, has shown potentials for consciousness rehabilitation of DOC patients as it is effective in regulating the central nervous system.

Methods and design: This protocol is a double-blind randomized sham-controlled crossover trial. Totally 30 participants will be randomly assigned to either group 1 or group 2 in a 1:1 ratio, with 15 patients in each group. Each patient will received 20 sessions, in which 10 sessions will be active and 10 will be sham, separated by 10-days washout period. The active-rTMS will include 10 Hz rTMS over the individual-targeted area on each participants. Primary and secondary evaluating indicators will be performed at each baseline and after rTMS treatment. Primary outcome will be determined as behavioral response to treatment as measured using the Coma Recovery Scale - Revised (CRS-R). Resting-state high-density EEG will be also recorded to investigate the neurophysiological correlates by rTMS.

Discussion:This study will contribute to define the role of rTMS for the treatment of DOC patients and characterise the neural correlates of its action. The investigators proposed a method of individualized target selection for DOC patients based on the existing gold standard CRS-R score and MRI, and used a cross randomized controlled trial to verify the role of rTMS in DOC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. acquired brain injuries less than 1 year and more than 28 days in DOC;
2. clinical diagnosis of DOC Disease;
3. no medical history of neuropsychiatric diseases;
4. no contraindications for rTMS or EEG, no sedatives in use or other drugs that might interfere with brain stimulation, such as Na+ or Ca2+ channel blockers or NMDA receptor antagonists;
5. stable state of disease and vital signs;
6. the families of the patients volunteered the patient to participate in the study and provided signed informed consent;
7. the integrity of the individualized stimulation target cortex are verified by MRI.

Exclusion Criteria:

1. patients in other non-invasive or invasive neuroregulation trials;
2. motor evoked potential (MEP) in M1 region cannot be induced by TMS pulse;
3. uncontrolled epilepsy, seizure within 4 weeks before enrollment;
4. metallic implant in the skull, pacemaker, craniotomy under the stimulated site, implanted brain device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline JFK Coma Recovery Scale-Revised(CRS-R) for Crossover Study 1 | immediately after 10 days individualized rTMS session
  The Coma Recovery Scale-Revised(CRS-R), a total of 23 points, is widely used to define the level of consciousness and assess neurobehavioral recovery of patients with DOC. It is based on six subscales that assess auditory(4 points), visual(5 points), motor(6 points), motor/speech(3 points), communication(2 points), and arousal processes(3 points). Each item of CRS-R is in good agreement with the diagnostic and differential diagnostic criteria of VS/UWS, MCS and EMCS. The higher scores mean a better outcome.
Change from Baseline JFK Coma Recovery Scale-Revised(CRS-R) for Crossover Study 2 | immediately after Washout period
  The Coma Recovery Scale-Revised(CRS-R), a total of 23 points, is widely used to define the level of consciousness and assess neurobehavioral recovery of patients with DOC. It is based on six subscales that assess auditory(4 points), visual(5 points), motor(6 points), motor/speech(3 points), communication(2 points), and arousal processes(3 points). Each item of CRS-R is in good agreement with the diagnostic and differential diagnostic criteria of VS/UWS, MCS and EMCS. The higher scores mean a better outcome.
Change from Baseline JFK Coma Recovery Scale-Revised(CRS-R) for Crossover Study 3 | immediately after 10 days sham rTMS session
  The Coma Recovery Scale-Revised(CRS-R), a total of 23 points, is widely used to define the level of consciousness and assess neurobehavioral recovery of patients with DOC. It is based on six subscales that assess auditory(4 points), visual(5 points), motor(6 points), motor/speech(3 points), communication(2 points), and arousal processes(3 points). Each item of CRS-R is in good agreement with the diagnostic and differential diagnostic criteria of VS/UWS, MCS and EMCS. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Resting-State EEG for Crossover Study 1 | immediately after 10 days individualized rTMS session
  EEG will be acquired from 66 channels with positions of the International 10-20 System for 10 mins. The relative spectral power (RSP) and functional connectivity (FC) of participants will be calculated by the selected artifact-free EEG epochs at five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz). The investigators will compute off-line analysis to calculate RSP and FC.
Change from Baseline Resting-State EEG for Crossover Study 2 | immediately after Washout period
  EEG will be acquired from 66 channels with positions of the International 10-20 System for 10 mins. The relative spectral power (RSP) and functional connectivity (FC) of participants will be calculated by the selected artifact-free EEG epochs at five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz). The investigators will compute off-line analysis to calculate RSP and FC.
Change from Baseline Resting-State EEG for Crossover Study 3 | immediately after 10 days sham rTMS session
  EEG will be acquired from 66 channels with positions of the International 10-20 System for 10 mins. The relative spectral power (RSP) and functional connectivity (FC) of participants will be calculated by the selected artifact-free EEG epochs at five frequency bands: δ (1-4 Hz), θ (4-8 Hz), α (8-13 Hz), β (13-30 Hz), and γ (30-45 Hz). The investigators will compute off-line analysis to calculate RSP and FC.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu C, Yuan Z, Chen Z, Liao Z, Li S, Feng Y, Tang Z, Nian J, Huang X, Zhong H, Xie Q. Perturbational complexity index in assessing responsiveness to rTMS treatment in patients with disorders of consciousness: a cross-over randomized controlled trial study. J Neuroeng Rehabil. 2024 Sep 19;21(1):167. doi: 10.1186/s12984-024-01455-1. PMID 39300529
- [Derived] Xu C, Zhu Z, Wu W, Zheng X, Zhong H, Huang X, Xie Q, Qian X. Effects of 10 Hz individualized repetitive transcranial magnetic stimulation on patients with disorders of consciousness: a study protocol for an exploratory double-blind crossover randomized sham-controlled trial. Trials. 2023 Apr 1;24(1):249. doi: 10.1186/s13063-023-07122-5. PMID 37005647
- [Derived] Xu C, Wu W, Zheng X, Liang Q, Huang X, Zhong H, Xiao Q, Lan Y, Bai Y, Xie Q. Repetitive transcranial magnetic stimulation over the posterior parietal cortex improves functional recovery in nonresponsive patients: A crossover, randomized, double-blind, sham-controlled study. Front Neurol. 2023 Feb 16;14:1059789. doi: 10.3389/fneur.2023.1059789. eCollection 2023. PMID 36873436

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05187000/Prot_000.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05187000/ICF_001.pdf